CLINICAL TRIAL: NCT02686593
Title: Clofarabine, Cytarabine and Mitoxantrone (CLAM) for Relapsed or Refractory AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOFAL07200
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Clofarabine; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine, AraC, mitoxantrone (CLAM) (Other): This is the single arm with the intervention using Clofarabine, AraC, Mitoxantrone
  Interventions: Drug: Clofarabine, AraC, mitoxantrone (CLAM)

INTERVENTIONS:
Drug: Clofarabine, AraC, mitoxantrone (CLAM) — The combination of clofarabine, cytarabine (Ara-C) and mitoxantrone will be used in patients with AML in first relapse or after failure of first salvage
  Other Names: CLAM

SUMMARY:
The study aims to evaluate the efficacy of the regimen CLAM in relapsed or refractory AML when used as first salvage for patients to relapse or fail after standard treatment with daunorubicin/cytarabine induction.

DETAILED DESCRIPTION:
Clofarabine, a second generation purine nucleoside analog, has been evaluated in several studies in relapsed AML.[1-3] Safety and dosages of clorafabine have already been determined in previous phase I/II studies. A demonstrable complete remission rate of up to 40% to 50% was shown in relapsed or refractory AML.[4-6] Since 2009, Clofarabine (40mg/m2/day for 5 days) in combination with high-dose cytarabine (2g/m2/day for 5 days) (CLARA) was adopted as the re-induction protocol for relapsed or refractory patients with AML at the Department of Medicine, Queen Mary Hospital. We have shown that this protocol is safe, tolerable and effective for relapsed AML. A recent updated analysis (Gill H et al., unpublished) showed a completed response rate of 50.8%. With the CLARA regimen, all patients (N=60) developed grade 3/4 neutropenia and thrombocytopenia. 8% developed grade 3/4 hepatotoxicity and 40% developed febrile neutropenia with clinical sepsis. There is increasing evidence to show that clofarabine is safe and efficacious when combined with the anthracyclines idarubicin or daunorubicin.7,8 In this prospective study, we combine clofarabine and cytarabine (Ara-C) with the topoisomerase II inhibitor mitoxantrone. In this protocol, the dosages of clofarabine and cytarabine will be reduced to 30mg/m2/day and 750mg/m2/day respectively, comparable to most clinical trials. In our previous publication of experience with the use of CLARA by Tse et al and Leung et al, clofarabine at 40mg/m2/day for 5 days was combined with high-dose cytarabine at 2g/m2/day.[5,6] The regimen was shown to be safe. The combination of clofarabine with anthracyclines has been evaluated. Mathiesen at al evaluated the CIA regimen comprising clofarabine at 20mg/m2/day from day 1 to day 5, idarubicin at 10mg/m2/day from day 1 to day 3 and cytarabine at 1g/m2/day from day 1 to day 5.[7] Abbie et al investigated the regimen comprising Clofarabine at 20mg/m2/day or 25mg/m2/day for 5 days in combination with mitoxantrone and etoposide.7 Based on the clinical trials and our extensive experience with the use of CLARA, the dosages of clofarabine in CLAM was determined. With the significant reduction in the dose of cytarabine to 750mg/m2/day for 5 days in CLAM, the dose of clofarabine was chosen at 30mg/m2/day for 5 days with the aim to maintain the efficacy seen with CLARA. The aim of this combination is to maintain or improve treatment efficacy seen with a lower treatment-related toxicity via dose reduction of clofarabine and cytarabine compared to CLARA. CLAM is expected to be safe and tolerable especially when used as first salvage in patient with a ECOG performance status of 0 or 1. The regimen CLAM has been approved by the institutional review board of Queen Mary Hospital/University of Hong Kong. In a pilot study, 4 patients used the regimen. 2 patients achieved a complete remission. Cardiotoxicity was not seen. Grade 3/4 hepatotoxicity was not seen. There were no treatment-related mortality observed. CLAM was shown to be safe and with manageable toxicity profile. In addition, less myeloid toxicity is expected during consolidation as patients who achieve a remission will have better marrow reserve when compared to those at relapse. Patients will have their cardiac, liver and renal function and performance status evaluated continuously and patients with cardiac dysfunction, significantly impaired renal or liver function and ECOG performance status of 2 or above will be excluded. Thus consolidation with the same dose as with induction is expected to be safe and tolerable.

The study aims to evaluate the efficacy of the regimen CLAM in relapsed or refractory AML when used as first salvage for patients to relapse or fail after standard treatment with daunorubicin/cytarabine induction. We aim to improve treatment efficacy at a more tolerable dose of clofarabine and cytarabine compared to CLARA.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory acute myeloid leukemia (AML) after one first-line chemotherapy regimen
2. Patients aged 18 - 65 inclusively
3. European Cooperative Oncology Group (ECOG) performance status of less than 2

Exclusion Criteria:

1. Patients aged less than 18 or above 65
2. ECOG performance status of 2 or more
3. Acute promyelocytic leukaemia
4. Uncontrolled active infection
5. Uncontrolled arrhythmia
6. Altered renal dysfunction with serum creatinine > 1.5 x ULN and/or creatinine clearance < 50 mL/min
7. Significant neurologic (grade > 2) or psychiatric disorder, dementia or seizures
8. Clinical symptoms suggesting active central nervous system leukemia
9. Severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock or disseminated intravascular coagulation
10. Patients with known HIV, Hepatitis B or C infection or history of cirrhosis
11. Patients Significant hepatic dysfunction: Direct bilirubin > 1.5 x upper limit of normal (ULN) for age; ALT or AST > 3 x upper limit of normal (ULN) for age; Lipase > 2.0 x upper limit of normal (ULN) for age
12. Females of childbearing potential must have a negative pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Response rate | Day 28
  Remission status will be assessed on day 28 of treatment for the assessment of response rate using standard criteria

SECONDARY OUTCOMES:
Leukemia-free survival | 2 years
  This is defined as time (in months) from remission after CLAM regimen to relapse (event), death (censor), HSCT (censor) or latest follow-up (censor).
Overall survival | 5 years
  This is defined as the time (in months) from recruitment to death (event) or latest follow-up (censor).
Adverse events | 1 year
  Toxicity will be defined using the NCI Common Terminology Criteria for Adverse Events (CTCAE). Data on all toxicities listed will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Singh, Harry Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faderl S, Gandhi V, Kantarjian HM. Potential role of novel nucleoside analogs in the treatment of acute myeloid leukemia. Curr Opin Hematol. 2008 Mar;15(2):101-7. doi: 10.1097/MOH.0b013e3282f46e94. PMID 18300755
- [Background] Faderl S, Ferrajoli A, Wierda W, Huang X, Verstovsek S, Ravandi F, Estrov Z, Borthakur G, Kwari M, Kantarjian HM. Clofarabine combinations as acute myeloid leukemia salvage therapy. Cancer. 2008 Oct 15;113(8):2090-6. doi: 10.1002/cncr.23816. PMID 18756533
- [Background] Sampat K, Kantarjian H, Borthakur G. Clofarabine: emerging role in leukemias. Expert Opin Investig Drugs. 2009 Oct;18(10):1559-64. doi: 10.1517/13543780903173222. PMID 19715446
- [Background] Becker PS, Kantarjian HM, Appelbaum FR, Petersdorf SH, Storer B, Pierce S, Shan J, Hendrie PC, Pagel JM, Shustov AR, Stirewalt DL, Faderl S, Harrington E, Estey EH. Clofarabine with high dose cytarabine and granulocyte colony-stimulating factor (G-CSF) priming for relapsed and refractory acute myeloid leukaemia. Br J Haematol. 2011 Oct;155(2):182-9. doi: 10.1111/j.1365-2141.2011.08831.x. Epub 2011 Aug 18. PMID 21848522
- [Background] Tse E, Leung AY, Sim J, Lee HK, Liu HS, Yip SF, Kwong YL. Clofarabine and high-dose cytosine arabinoside in the treatment of refractory or relapsed acute myeloid leukaemia. Ann Hematol. 2011 Nov;90(11):1277-81. doi: 10.1007/s00277-011-1223-2. Epub 2011 Apr 1. PMID 21455604
- [Background] Leung AY, Tse E, Hwang YY, Chan TS, Gill H, Chim CS, Lie AK, Kwong YL. Primary treatment of leukemia relapses after allogeneic hematopoietic stem cell transplantation with reduced-intensity conditioning second transplantation from the original donor. Am J Hematol. 2013 Jun;88(6):485-91. doi: 10.1002/ajh.23439. Epub 2013 May 2. PMID 23512868
- [Background] Nazha A, Kantarjian H, Ravandi F, Huang X, Choi S, Garcia-Manero G, Jabbour E, Borthakur G, Kadia T, Konopleva M, Cortes J, Ferrajoli A, Kornblau S, Daver N, Pemmaraju N, Andreeff M, Estrov Z, Du M, Brandt M, Faderl S. Clofarabine, idarubicin, and cytarabine (CIA) as frontline therapy for patients </=60 years with newly diagnosed acute myeloid leukemia. Am J Hematol. 2013 Nov;88(11):961-6. doi: 10.1002/ajh.23544. Epub 2013 Sep 9. PMID 23877926
- [Background] Vigil CE, Tan W, Deeb G, Sait SN, Block AW, Starostik P, Griffiths EA, Thompson JE, Greene JD, Ford LA, Wang ES, Wetzler M. Phase II trial of clofarabine and daunorubicin as induction therapy for acute myeloid leukemia patients greater than or equal to 60 years of age. Leuk Res. 2013 Nov;37(11):1468-71. doi: 10.1016/j.leukres.2013.07.036. Epub 2013 Aug 15. PMID 24011826
- [Background] Abbi KK, Rybka W, Ehmann WC, Claxton DF. Phase I/II study of clofarabine, etoposide, and mitoxantrone in patients with refractory or relapsed acute leukemia. Clin Lymphoma Myeloma Leuk. 2015 Jan;15(1):41-6. doi: 10.1016/j.clml.2014.06.005. Epub 2014 Jun 11. PMID 25085441
- [Derived] Gill H, Yim R, Pang HH, Lee P, Chan TSY, Hwang YY, Leung GMK, Ip HW, Leung RYY, Yip SF, Kho B, Lee HKK, Mak V, Chan CC, Lau JSM, Lau CK, Lin SY, Wong RSM, Li W, Ma ESK, Li J, Panagiotou G, Sim JPY, Lie AKW, Kwong YL. Clofarabine, cytarabine, and mitoxantrone in refractory/relapsed acute myeloid leukemia: High response rates and effective bridge to allogeneic hematopoietic stem cell transplantation. Cancer Med. 2020 May;9(10):3371-3382. doi: 10.1002/cam4.2865. Epub 2020 Mar 18. PMID 32187883